CLINICAL TRIAL: NCT05452109
Title: Improvement of Football-Related Performance Parameters: Application of Blood Flow Restrictive Exercise
Brief Title: Effect of Blood Flow Restriction on Football-Related Performance Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DrTez
Record Dates: First submitted 2022-06-01; First posted 2022-07-11 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-06

CONDITIONS: Vascular Occlusion; Soccer; Exercise; EMG
MeSH Terms: conditions — Motor Activity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction + Classical Training (Experimental)
  Interventions: Other: Blood Flow Restriction
- Classical Training Alone (Experimental)
  Interventions: Other: Classical Training Alone

INTERVENTIONS:
Other: Blood Flow Restriction — Blood flow restriction with low load (30-50% 1RM) for 2 sessions in a week for 6 weeks during classical training will be applied.
  Arms: Blood Flow Restriction + Classical Training
Other: Classical Training Alone — Classical training same as Group 1with moderate to high load (70-90% 1RM) for 2 sessions in a week for 6 weeks will be applied without blood restriction.
  Arms: Classical Training Alone

SUMMARY:
The blood flow restriction method can have similar or superior effects to high-intensity exercises even in a short duration, which can positively affect some performance parameters, can be applied with low-intensity load and cause hypertrophy in the muscle by providing high metabolic stress, facilitating muscle growth without significantly changing the total training dose. The aim of this study is to investigate whether adding the blood flow restriction method to the classical training program can be more effective than the classical training applied alone in the development of football-related performance parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being a male between the ages of 18-30 years
* Volunteer to participate in the study
* Playing football in one of the clubs in Istanbul for at least 1 year
* Being in the pre-season of the club
* Absence of any ongoing musculoskeletal problems that limit exercising

Exclusion Criteria:

* Having at least one of the contraindications preventing the application of blood flow restriction (Smoking, previous venous thromboembolism, risk of peripheral vascular disease (ankle-brachial index <0.9), coronary heart disease, hypertension, hemophilia, etc.).
* History of sports injury in the last 6 months
* Orthopedic lower extremity surgery in the last 1 year
* Body mass index ≥ 30 kg/m2

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of Muscle Strength and Endurance | 6 weeks
  Isokinetic dynamometer

SECONDARY OUTCOMES:
Evaluation of Lower Extremity Power | 6 weeks
  Vertical jump test
Evaluation of Aerobic Endurance | 6 weeks
  Yo-Yo Intermittent Recovery Level 1 test
Evaluation of Change of Direction Speed | 6 weeks
  T Test
Evaluation of Reactive Agility | 6 weeks
  Y-Shaped Reactive Agility Test
Evaluation of Dynamic Balance | 6 weeks
  Y Balance Test
Systemic Fatigue | 6 weeks
  Lactate analysis
General Perceived Fatigue | 6 weeks
  Borg scale
Evaluation of General Satisfaction and Perceived Performance Change | 6th week
  General satisfaction and the change in performance perceived by the participants will be evaluated with the 7 points Global Rating of Change Scale after the training program. According to the scale, it is expressed as "-3: I am much worse, -2: I am worse, -1: I am a little worse, 0: No change, 1: I am a little better, 2: I am better, 3: I am much better".

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpözgen, PhD, Study Chair — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Biruni University, Istanbul
  - Istanbul University Cerrahpasa, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kara Kaya B, Alpozgen AZ, Alpozgen MR, Dikmen G. Performance and injury-related effects of low-load blood flow restriction training in amateur soccer players: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Dec 20. doi: 10.1186/s13102-025-01416-8. Online ahead of print. PMID 41422254